CLINICAL TRIAL: NCT03426748
Title: A Phase III Randomized Study of Low Dose Rate Compared to High Dose Rate Prostate Brachytherapy for Favorable Risk and Low Tier Intermediate Risk Prostate Cancer
Brief Title: LDR vs. HDR Brachytherapy for Prostate Cancer
Acronym: LDR/HDRmono
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: BC Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H17-02904
Record Dates: First submitted 2018-02-02; First posted 2018-02-08 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: Brachytherapy; Quality of life; High dose rate vs. low dose rate; Intermediate risk group
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low dose rate brachytherapy (Active Comparator): Device: Radiation. Low dose rate prostate brachytherapy is delivered under anesthesia in a single 1.5-2 hour procedure as an out-patient. The men return 4 weeks later for detailed imaging to assess implant quality.
  Interventions: Radiation: Low dose rate prostate brachytherapy
- High dose rate brachytherapy (Experimental): Device: Radiation. High dose rate prostate brachytherapy is delivered in 2 procedures, 2 weeks apart, also under anesthesia, but no follow-up imaging visit is required.
  HDR brachytherapy is also accomplished as an out-patient.
  Interventions: Radiation: High dose rate prostate brachytherapy

INTERVENTIONS:
Radiation: Low dose rate prostate brachytherapy — Permanent implantation of radioactive Iodine-125 seeds under anesthesia with ultrasound guidance
  Other Names: permanent seed implant
  Arms: Low dose rate brachytherapy
Radiation: High dose rate prostate brachytherapy — Temporary implantation of radioactive material into the prostate in the form of a stepping source of Iridium 192 that travels through 16-18 needles or catheters strategically placed through the prostate
  Other Names: HDR brachytherapy
  Arms: High dose rate brachytherapy

SUMMARY:
H17-02904 is a randomized comparison of low dose rate vs. high dose rate prostate brachytherapy for favorable and intermediate risk prostate cancer suitable for brachytherapy as monotherapy. This is a continuation with expanded accrual of the randomized Pilot study H15-02103

DETAILED DESCRIPTION:
Men suitable for prostate brachytherapy as monotherapy will undergo multiparametric Magnetic Resonance Imaging for staging and identification of a dominant lesion and will be randomly selected for either a single low dose rate permanent seed implant or 2 fractions of high dose rate brachytherapy. Using image registration techniques, dominant lesions will be biopsied under anesthesia at the start of the brachytherapy procedure. Biopsies will reviewed for tumor Gleason score and sent for Cell Cycle Progression testing (Prolaris). Patients receiving high dose rate brachytherapy will also have biopsies between the 2 fractions to assess tumor changes induced from the first fraction. Post implant quality assurance will determine the dose to the dominant lesions and compare these between the 2 types of brachytherapy. Post implant symptoms will be tracked for severity and time course.

ELIGIBILITY:
Inclusion Criteria:

Favorable risk and low-tier intermediate-risk prostate cancer with estimated life expectancy of at least 10 years.

* Clinical stage T1c-T2b, PSA < 20, Gleason < 8
* ECOG 0-1
* Low tier intermediate-risk prostate cancer is defined by a single NCCN intermediate risk factor
* Extensive favorable-risk disease is defined as:

  * clinical stage T1c-T2a
  * PSA < 10
  * Gleason 6
  * ≥ 50% of biopsy cores containing cancer
  * PSA density > 0.2 ng/cc
* Selected intermediate risk patients not defined above

  * - T1c/T2a
  * - PSA < 10
  * -Gleason 4+3
  * PSA > 10 and Gleason 3+4
  * PSA 10-15 ng/ml and Gleason 4+3
  * -< 33% of cores involved
  * -Max tumor length in any core 10 mm
* No androgen deprivation therapy (ADT)
* Prostate volume by TRUS ≤ 60 cc.
* Not eligible for, or accepting of, active surveillance according to NCCN guidelines.
* Signed study specific informed consent.

Exclusion Criteria:

* Prior radical surgery for carcinoma of the prostate,
* Prior pelvic radiation
* Prior chemotherapy for prostate cancer,
* Prior TURP or cryosurgery of the prostate
* Claustrophobic or unable to undergo MRI

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2034-10-31 (Estimated)

PRIMARY OUTCOMES:
The difference in Quality of Life in the urinary domain between LDR and HDR brachytherapy. | 0-60 months
  The urinary domain of the EPIC prostate cancer specific QOL questionnaire will be assessed.

SECONDARY OUTCOMES:
Quality of Life in the bowel and sexual domains | 0-60 months
  The EPIC score in the bowel and sexual domains will be evaluated at baseline, 1, 3, 6, 12, 24, 36, 48 and 60 months
Time to return to baseline +/- 3 points for the International Prostate Symptom Score | 0-60 months
  The IPS Score will be assessed at baseline, 1, 3, 6, 12, 24, 36, 48 and 60 months
Acute and long term toxicity | [Time Frame: 0-10 years]
  Acute and long-term toxicity will be graded using the Common Terminology Criteria for Adverse Events (CTCAE V4) at each follow up time point
Biochemical Outcome | 5-10 years
  PSA will be recorded every 6 months to 5 years and then annually to 10 years
Histologic Outcome | 3 years
  Prostate re-biopsy will be performed at 36 months to assess the local efficacy of treatment
Cell cycle progression score | 1 month to 10 years
  For those patients consenting to targeted biopsies under anesthesia at the start of their brachytherapy procedure (separate optional consent) MRI-TRUS fusion accuracy will be verified by targeted biopsies and Biopsy material will be sent for genetic testing to determine Cell cycle Progression scores for both arms of the trial to ultimately correlate with outcome.
Tumor oxygenation and cell cycle distribution | 1 month to 10 years.
  For patients receiving 2 fractions of high dose rate brachytherapy, biopsy between the 2 fractions will assess radiosensitivity by evaluating changes in oxygenation and cell cycle distribution between the 2 fractions, for ultimate correlation with efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Ross Halperin, MD, Study Director — British Columbia Cancer Agency Program Director
Locations (1):
- British Columbia Cancer Agency Center for the Southern Interior, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crook J, Ots A, Gaztanaga M, Schmid M, Araujo C, Hilts M, Batchelar D, Parker B, Bachand F, Milette MP. Ultrasound-planned high-dose-rate prostate brachytherapy: dose painting to the dominant intraprostatic lesion. Brachytherapy. 2014 Sep-Oct;13(5):433-41. doi: 10.1016/j.brachy.2014.05.006. Epub 2014 Jun 20. PMID 24958556
- [Background] Batchelar D, Gaztanaga M, Schmid M, Araujo C, Bachand F, Crook J. Validation study of ultrasound-based high-dose-rate prostate brachytherapy planning compared with CT-based planning. Brachytherapy. 2014 Jan-Feb;13(1):75-9. doi: 10.1016/j.brachy.2013.08.004. Epub 2013 Sep 27. PMID 24080299
- [Background] Schmid M, Crook JM, Batchelar D, Araujo C, Petrik D, Kim D, Halperin R. A phantom study to assess accuracy of needle identification in real-time planning of ultrasound-guided high-dose-rate prostate implants. Brachytherapy. 2013 Jan-Feb;12(1):56-64. doi: 10.1016/j.brachy.2012.03.002. Epub 2012 Apr 17. PMID 22513104

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-07): https://cdn.clinicaltrials.gov/large-docs/48/NCT03426748/Prot_SAP_000.pdf